CLINICAL TRIAL: NCT01086436
Title: Reactogenicity and Safety of a Single Dose of GlaxoSmithKline (GSK) Biologicals' Human Rotavirus (HRV) Vaccine (444563) in Healthy Children
Brief Title: Study to Evaluate the Safety of Rotarix™ in Chinese Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113552
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Infections, Rotavirus
Keywords: Human Rotavirus vaccine
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rotavirus Group (Experimental): Subjects will receive Rotarix™
  Interventions: Biological: Rotarix ™
- Placebo Group (Placebo Comparator): Subjects will receive placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix ™ — Oral, single dose
  Arms: Rotavirus Group
Biological: Placebo — Oral, single dose
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to assess the safety of Rotarix ™ when administered in healthy children aged 2 to 6 years in China.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians (Legally acceptable representative) can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female subject of Chinese origin, between, and including, 2 and 6 years of age at the time of vaccination.
* Written informed consent obtained from the parent or legally acceptable representative of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs six months prior to the vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 14 days of the Human Rotavirus vaccine or placebo with the exception of the routine childhood vaccines. Routine childhood vaccines must not be administered on the same day as the Human Rotavirus vaccine or placebo.
* Administration of immunoglobulins and/or any blood products since birth within three months preceding the study vaccine or planned administration during the study period.
* Major congenital defects or serious chronic illness.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of Intusussception or any chronic gastrointestinal disease that would predispose for Intusussception including any uncorrected congenital malformation of the gastrointestinal tract.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Gastroenteritis within 7 days preceding the study vaccine or placebo administration.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product..
* Child in care.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-03-13 (Actual); Primary Completion 2010-04-16 (Actual); Study Completion 2010-04-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of each solicited symptom | Within the 8-day (Day 0 - Day 7) follow-up period after the vaccine dose.

SECONDARY OUTCOMES:
Occurrence of unsolicited adverse events | Within the 31 days (Day 0 - Day 30) after the vaccine dose.
Occurrence of serious adverse events | Throughout the study period following the vaccine dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Liucheng County, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Li RC, Li YP, Mo ZJ, Luo D, Huang T, Kong JL, Wang LH, Song NS, Liu A, Zhang H, Liao X, Karkada N, Han HH. Reactogenicity and safety of a liquid human rotavirus vaccine (RIX4414) in healthy adults, children and infants in China: randomized, double-blind, placebo-controlled Phase I studies. Hum Vaccin Immunother. 2013 Aug;9(8):1638-42. doi: 10.4161/hv.25076. Epub 2013 Jun 4. PMID 23807360
- See also: Results for study 113552 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/113552?search=study&b%22b''%22#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register